CLINICAL TRIAL: NCT06508151
Title: Study on the Effectiveness and Safety of Neovaginoplasty Using Photoinduced-imine-crosslink Hydrogel in Patients With Mayer-Rokitansky-Kuster-Hauser Syndrome
Brief Title: Neovaginoplasty Using Photoinduced-imine-crosslink Hydrogel in MRKH Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Obstetrics & Gynecology Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Keqin Hua, Doctor, Principal Investigator, Clinical Professor, Obstetrics & Gynecology Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-16
Record Dates: First submitted 2024-06-27; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Mayer Rokitansky Kuster Hauser Syndrome
Keywords: Photoinduced-imine-crosslink hydrogel; MRKH syndrome; Neovaginoplasty
MeSH Terms: conditions — Mullerian aplasia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): After neovaginoplasty, a vaginal mold spreaded with photoinduced-imine-crosslink hydrogel was placed in the neovagina.
  Interventions: Procedure: neovaginoplasty and vaginal mold spreaded with photoinduced-imine-crosslink hydrogel
- Arm 2 (Other): After neovaginoplasty, a vaginal mold was placed in the neovagina directly without anything spreaded.
  Interventions: Procedure: neovaginoplasty and vaginal mold

INTERVENTIONS:
Procedure: neovaginoplasty and vaginal mold spreaded with photoinduced-imine-crosslink hydrogel — Under general anesthesia and catheterized bladder, the patient was in the lithotomy position. In the connective tissue plane between the bladder and rectum, the vestiges of the müllerian ducts were identified. With the index finger in the rectum as a direction and protection, Hegar's dilators of increasing size (4.5-10) were pushed through the dimples gently. After that, a double-barreled canal appeared. Then, the raphe between the canals was incised. The neovagina was created. According to the randomization, a vaginal mold spreaded with hydrogel or not was placed in the neovagina for 6 months. The patients were suggested to wear the vaginal mold continuously over the following 6 months. After that, they were allowed to have the first sexual intercourse. Otherwise, the mold wearing time was 1 h daily, until they had sexual activity at least twice a week.
  Arms: Arm 1
Procedure: neovaginoplasty and vaginal mold — Under general anesthesia and catheterized bladder, the patient was in the lithotomy position. In the connective tissue plane between the bladder and rectum, the vestiges of the müllerian ducts were identified. With the index finger in the rectum as a direction and protection, Hegar's dilators of increasing size (4.5-10) were pushed through the dimples gently. After that, a double-barreled canal appeared. Then, the raphe between the canals was incised. The neovagina was created. According to the randomization, a vaginal mold spreaded with hydrogel or not was placed in the neovagina for 6 months. The patients were suggested to wear the vaginal mold continuously over the following 6 months. After that, they were allowed to have the first sexual intercourse. Otherwise, the mold wearing time was 1 h daily, until they had sexual activity at least twice a week.
  Arms: Arm 2

SUMMARY:
Evaluating the effectiveness and safety of neovaginoplasty using photoinduced-imine-crosslink hydrogel in patients with MRKH syndrome by comparing the differences in the degree of squamous epithelialization, vaginal length and width, and sexual life quality.

DETAILED DESCRIPTION:
This is a randomized controlled trial. Patients meeting the inclusion criteria will be enrolled in this study: 1)Diagnosed with MRKH syndrome; 2)Without previous treatments; 3)Age: 18-35 years old; 4)Voluntary agreement to participate in the study, sign the informed consent form, and demonstrate good compliance with follow-up.

A centralized block randomization will be used to randomly assign patients to ensure that there will be an equal number of patients (1:1) in the hydrogel group and control group. The sample size is 20.

Under general anesthesia and catheterized bladder, the patient was in the lithotomy position. In the connective tissue plane between the bladder and rectum, the vestiges of the müllerian ducts were identified. With the index finger in the rectum as a direction and protection, Hegar's dilators of increasing size (4.5-10) were pushed through the dimples gently. After that, a double-barreled canal appeared. Then, the raphe between the canals was incised. The neovagina was created. According to the randomization, a vaginal mold spreaded with hydrogel or not was placed. The patients were suggested to wear the vaginal mold continuously over the following 6 months. After that, they were allowed to have the first sexual intercourse. Otherwise, the mold wearing time was 1 h daily, until they had sexual activity at least twice a week.

The primary endpoint is the degree of vaginal squamous epithelialization 1 month, 3 months, 6 months after surgery. The secondary endpoints include neovaginal length and width, sexual life quality, and surgical complications.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with MRKH syndrome;
2. Without previous related treatments; 3)18-35 years old;

4)Voluntary agreement to participate in the study, sign the informed consent form, and demonstrate good compliance with follow-up.

Exclusion Criteria:

1. With any previous artificial colpoplasty or other related treatment;
2. With history of diabetes or systemic immune system disease.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Degree of vaginal squamous epithelialization | 1 month
  Percentage of squamous epithelialization of neovagina
Degree of vaginal squamous epithelialization | 3 months
  Percentage of squamous epithelialization of neovagina
Degree of vaginal squamous epithelialization | 6 months
  Percentage of squamous epithelialization of neovagina

SECONDARY OUTCOMES:
length of neovagina | 1 month
  length in centimetre, measured by a ruler
length of neovagina | 3 months
  length in centimetre, measured by a ruler
length of neovagina | 6 months
  length in centimetre, measured by a ruler
width of neovagina | 1 month
  width in centimetre, measured by ruler
width of neovagina | 3 months
  width in centimetre, measured by ruler
width of neovagina | 6 months
  width in centimetre, measured by ruler
Sexual life quality | 6 months
  Female Sexual Function Index, a self-reported questionnaire to measure sexual life quality
Sexual life quality | 1 year
  Female Sexual Function Index, a self-reported questionnaire to measure sexual life quality

CONTACTS AND LOCATIONS:
Overall Officials: Keqin Hua, Doctor, Principal Investigator — Obstetrics & Gynecology Hospital of Fudan University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhang X, Qiu J, Ding J, Hua K. Comparison of neovaginoplasty using acellular porcine small intestinal submucosa graft or Interceed in patients with Mayer-Rokitansky-Kuster-Hauser syndrome. Arch Gynecol Obstet. 2019 Dec;300(6):1633-1636. doi: 10.1007/s00404-019-05352-0. Epub 2019 Oct 30. PMID 31667605
- [Result] Bao B, Zeng Q, Li K, Wen J, Zhang Y, Zheng Y, Zhou R, Shi C, Chen T, Xiao C, Chen B, Wang T, Yu K, Sun Y, Lin Q, He Y, Tu S, Zhu L. Rapid fabrication of physically robust hydrogels. Nat Mater. 2023 Oct;22(10):1253-1260. doi: 10.1038/s41563-023-01648-4. Epub 2023 Aug 21. PMID 37604908
- [Result] Zhang W, Bao B, Jiang F, Zhang Y, Zhou R, Lu Y, Lin S, Lin Q, Jiang X, Zhu L. Promoting Oral Mucosal Wound Healing with a Hydrogel Adhesive Based on a Phototriggered S-Nitrosylation Coupling Reaction. Adv Mater. 2021 Dec;33(48):e2105667. doi: 10.1002/adma.202105667. Epub 2021 Oct 4. PMID 34605063
- [Result] Hong Y, Zhou F, Hua Y, Zhang X, Ni C, Pan D, Zhang Y, Jiang D, Yang L, Lin Q, Zou Y, Yu D, Arnot DE, Zou X, Zhu L, Zhang S, Ouyang H. A strongly adhesive hemostatic hydrogel for the repair of arterial and heart bleeds. Nat Commun. 2019 May 14;10(1):2060. doi: 10.1038/s41467-019-10004-7. PMID 31089131